CLINICAL TRIAL: NCT00361296
Title: K562/GM-CSF Vaccination in Patients With Myelodysplastic Syndrome
Brief Title: Vaccine Therapy in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Alliance for Cancer Gene Therapy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J05115; P30CA006973 (NIH); NA_00001530 (Other: JHMIRB)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; refractory cytopenia with multilineage dysplasia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- K562/GM-CSF cell vaccine (Experimental): Vaccinations of 1x10^8 cells are given to participants at weeks 0, 3, 6, 9, and 17.
  Interventions: Biological: K562/GM-CSF cell vaccine

INTERVENTIONS:
Biological: K562/GM-CSF cell vaccine

SUMMARY:
RATIONALE: Vaccines made from cancer cells may help the body build an effective immune response to kill abnormal cells.

PURPOSE: This clinical trial is studying how well vaccine therapy works in treating patients with myelodysplastic syndromes (MDS).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of GM-K562 cell vaccine in patients with myelodysplastic syndromes.
* Determine the hematologic and cytogenetic response in patients treated with this vaccine.

Secondary

* Determine if vaccination with GM-K562 cell vaccine can induce an immune response to common myeloid antigens (e.g., Wilms' tumor-1 [WT-1], survivin, or proteinase-3), as defined by a 30% increase from baseline in specific cytotoxic T-cells measured by Elispot assay, in patients with myelodysplastic syndromes.
* Determine if immune response correlates with any clinical responses (e.g., hematologic response, resolution of cytogenetic abnormalities, or decrease in other parameters, such as WT-1 mRNA levels).

OUTLINE: This is an open-label study.

Patients receive GM-K562 cell vaccine subcutaneously once in weeks 0, 3, 6, 9, and 17 in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples are collected periodically for correlative and biomarker studies. Samples are analyzed by cytogenetic studies, fluorescent in situ hybridization (FISH), and flow cytometry. Elispot is used to quantify cellular cytotoxic T-cell response to Wilms' tumor-1 (WT-1), survivin, and proteinase 3.

After completion of study treatment, patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed myelodysplastic syndromes (MDS), including any of the following:

  * Refractory anemia (RA)
  * RA with ringed sideroblasts
  * Refractory cytopenias with multilineage dysplasia (RCMD)
  * RCMD with ringed sideroblasts
  * RA with excess blasts 1 (5-9% blasts)
  * RA with excess blasts 2 (10-19% blasts)
* Must have poor-risk MDS, defined by the following:

  * At least 2 lineages involved
  * Unfavorable cytogenetics (i.e., abnormalities of chromosome 5 or 7, 11q23, t[6;9], trisomy 8, inv3, or multiple/complex karyotype)
  * Transfusion requirement of > 2 units of packed red blood cells monthly
* No chronic myelomonocytic leukemia
* No transformation to acute myeloid leukemia

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine < 2.5 mg/dL
* Bilirubin < 2.5 mg/dL (unless due to Gilbert's syndrome)
* Room air oxygen saturation ≥ 94% at rest
* Fertile patients must use effective contraception
* Negative pregnancy test
* No other malignancy within the past 5 years except in situ cervical cancer or adequately treated nonmelanoma skin cancer
* No active autoimmune disease or history of autoimmune disease requiring systemic immunosuppressants including, but not limited to, any of the following:

  * Autoimmune hemolytic anemia
  * Idiopathic thrombocytopenia purpura
  * Inflammatory bowel disease
  * Vasculitis
  * Thyroiditis
  * Rheumatic illnesses
* No known HIV serum antibody positivity
* No other disease requiring long-term corticosteroids or other immunosuppressants, such as severe chronic obstructive pulmonary disease or asthma

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior systemic corticosteroids or other immunosuppressants (e.g., cyclosporine, azathioprine, tacrolimus, or mycophenolate mofetil)
* At least 3 weeks since prior growth factors
* At least 2 months since prior azacitidine for MDS
* No prior bone marrow or other organ transplantation
* No concurrent cytotoxic-based therapy for MDS
* No other concurrent growth factors, including epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Douglas Smith, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robinson TM, Prince GT, Thoburn C, Warlick E, Ferguson A, Kasamon YL, Borrello IM, Hess A, Smith BD. Pilot trial of K562/GM-CSF whole-cell vaccination in MDS patients. Leuk Lymphoma. 2018 Dec;59(12):2801-2811. doi: 10.1080/10428194.2018.1443449. Epub 2018 Apr 4. PMID 29616857

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were screen failures. 2 additional participants were removed from study by physician decision prior to receiving protocol intervention, so they never started the study.
Groups:
- K562/GM-CSF Cell Vaccine: Vaccinations of 1x10^8 cells are given to participants at weeks 0, 3, 6, 9, and 17.
  K562/GM-CSF cell vaccine
Period: Overall Study
Arm/Group | K562/GM-CSF Cell Vaccine
Started | 5
Completed | 2
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | K562/GM-CSF Cell Vaccine
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 64 [55 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response Rate as Assessed by Number of Participants Achieving a Major Hematologic Response
Description: A major hematologic response is defined as any of the following: hemoglobin increase >= 2 g/dL from baseline; platelet increase >= 30k/mcL from baseline; or neutrophil increase >= 100% or >= 500/mcL from baseline.
Time Frame: Baseline, week 21 post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | K562/GM-CSF Cell Vaccine
Number analyzed (Participants) | 5
Participants | 1

2. Primary Outcome: Cytogenetic Response Rate as Assessed by Number of Participants Achieving a Cytogenetic Response
Description: Cytogenetic response is defined as normalization of pretreatment cytogenetic abnormalities.
Time Frame: Week 21
Measure: Count of Participants; unit: Participants
Arm/Group | K562/GM-CSF Cell Vaccine
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Immune Response Rate as Assessed by Number of Participants Who Exhibit Induced Immune Response to WT-1, Survivin, or Proteinase-3
Description: Immune response to WT-1, survivin, or proteinase-3 as defined by a 30% increase from baseline in cytotoxic T cells measured by Elispot analysis.
Time Frame: Baseline, week 21 post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | K562/GM-CSF Cell Vaccine
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Combined Immune and Clinical Response Rate
Description: Number of participants who exhibited both an immune response as defined by Outcome 3 and a hematologic or cytogenetic response as defined by Outcomes 1 and 2, respectively.
Time Frame: Week 21 post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | K562/GM-CSF Cell Vaccine
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: Adverse events were collected at weeks 3, 6, 9, 13, 17, and every three months after week 21 for a total of one additional year.
Arm/Group | K562/GM-CSF Cell Vaccine
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | K562/GM-CSF Cell Vaccine (N=5)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Adenopathy (Immune system disorders) | 2 (2)
ALT elevated (Investigations) | 2 (2)
Altered mental status (Nervous system disorders) | 1 (1)
Anemia (Investigations) | 1 (2)
Anorexia (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
AST elevated (Investigations) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Bleeding - eye (Eye disorders) | 1 (1)
Bruising (General disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine elevated (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (Cardiac disorders) | 3 (5)
Erythema - mouth (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (3)
Flushing (General disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 4 (6)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Hyperphosphatemia (Investigations) | 1 (1)
Hyperuricemia (Investigations) | 1 (1)
Injection site reactions (Immune system disorders) | 5 (25)
Insomnia (General disorders) | 2 (2)
Leukopenia (Investigations) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Neuropathy (Nervous system disorders) | 2 (2)
Neutropenia (Investigations) | 1 (1)
Epistaxis (General disorders) | 1 (1)
Pain - flank (Musculoskeletal and connective tissue disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Respiratory infection (Infections and infestations) | 2 (3)
Sore throat (General disorders) | 1 (1)
Swollen gums (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Taste changes (Nervous system disorders) | 1 (2)
Thrombocytopenia (Investigations) | 2 (4)
Tinnitus (Nervous system disorders) | 1 (1)
Transfusion reaction (Immune system disorders) | 1 (2)
Vision changes (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)
Xerophthalmia (Eye disorders) | 1 (1)
Xerosis (Skin and subcutaneous tissue disorders) | 1 (1)
Zoster infection (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes